CLINICAL TRIAL: NCT04962360
Title: The Effect of Nutritional Formula Supplementation on Linear Growth of GH Treated Prepubertal Children With Idiopathic Short Stature (ISS) After 2 Years From the Beginning of GH-therapy: a Randomized, Double- Blind, Placebo-controlled Trial
Brief Title: The Effect of Nutritional Formula Supplementation on Linear Growth of Growth Hormone (GH) Treated Prepubertal Children With Idiopathic Short Stature (ISS) After 2 Years From the Beginning of GH-therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc26021ctil
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: ISS- Idiopathic Short Stature

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional standardized supplementation formula. (Experimental): Powder added to water, containing about 25% of recommended daily recommended intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake.
  Interventions: Dietary Supplement: Nutritional supplementation standardized formula
- Placebo (Placebo Comparator): Low caloric formula (Powder added to water) without added vitamins and minerals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation standardized formula — Powder added to water, containing about 25% of recommended Daily Recommended Intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake
  Arms: Nutritional standardized supplementation formula.
Dietary Supplement: Placebo — Low caloric formula (Powder added to water) without added vitamins and minerals
  Arms: Placebo

SUMMARY:
The proposed study is a double blind, randomized, placebo controlled study. The aim of the study is to evaluate the effect of combined growth hormone (GH) treatment &nutritional formula supplementation versus GH & placebo on growth parameters in 64 children with Idiopathic Short Stature (ISS) after the second year of GH treatment.

Participants will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1. Both participants and study team will be blinded to the type of treatment that each patient will receive during the study. The randomization will be done according to gender.

Participants in the intervention groups will be treated with the study formula and participants in the control group will be treated with a placebo low caloric formula (powder added to water). The study will continue for 6 months of intervention versus active placebo, with additional 6 months (an extension period), in which participants at both groups, the intervention and the placebo, will be offered to continue their participation in the study with the active study supplement.

ELIGIBILITY:
Inclusion Criteria:

1. GH treatment for at least 24 months due to idiopathic short stature (ISS)
2. Age 5-10 years inclusive.
3. Tanner stage 1 (gonadarche).
4. BMI <85 percentile for age and gender.

Exclusion Criteria:

1. SGA/ IUGR
2. Diagnosis of GH deficiency
3. Any known morbidity: chronic disease dysmorphic syndromes, bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardial, renal or pulmonary problems, metabolic disorders.
4. Any known gastrointestinal problem including absorption problems.
5. Any chronic treatment with medication that might affect appetite, weight or growth (for example SSRI's, steroids).
6. Any eating disorders and/or psychiatric disorder
7. Milk or other food allergies

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
height standard deviation score (SDS) | at 6 moths
weight standard deviation score | at 6 months

SECONDARY OUTCOMES:
BMI SDS | at 6 months
Lean body mass | at 6 months
muscle mass | at 6 months
Fat mass | at 6 months
Fat mass percentage | at 6 months

OTHER OUTCOMES:
height SDS | at 12 months
Weight SDS | at 12 months
BMI SDS | at 12 months
Lean body mass | at 12 months
muscle mass | at 12 months
fat mass | at 12 months
fat mass percentage | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schnieder Children's Medical Center
Locations (1):
- Schneider children's medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No